CLINICAL TRIAL: NCT00607269
Title: Voucher-Based Incentives in a Prevention Setting
Acronym: VIPS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIDA 015990; R01DA015990 (NIH)
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Results first posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Substance-related Disorders
Keywords: Drug Abuse; Contingency management; Voucher-based Reinforcement Therapy; Homosexuality; Homeless Persons
MeSH Terms: conditions — Substance-Related Disorders; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control condition receiving minimal incentives for service program attendance and participation.
- Contingency Management (Experimental): Contingency management (Voucher-Based Reinforcement Therapy) intervention providing positive reinforcement for service program participation and attendance, enactment of prosocial/health behavior, and/or clean urine samples (i.e., no illicit drug use) and clean breathalyzer tests (i.e., BA < 0.05).
  Interventions: Behavioral: Voucher-Based Reinforcement Therapy

INTERVENTIONS:
Behavioral: Voucher-Based Reinforcement Therapy — Participants were randomized into either the CM or control condition. Both conditions earned points for attendance and participation (max 364 points).
  Participants in the CM condition also earned points for targeted health-promoting behaviors and for drug/alcohol abstinence. CM points for targeted health-promoting behaviors were not limited. Points for abstaining from substance use were awarded based on a Level 1 (recent abstinence for amphetamine, methamphetamine, PCP, and cocaine metabolites, as well as blood alcohol <0.05) urine sample.
  Other Names: VIPS
  Arms: Contingency Management

SUMMARY:
This study evaluates a contingency management program that rewards homeless, non-treatment-seeking substance abusing men who have sex with men (MSM) for abstaining from drugs and for performing prosocial behaviors. If this program motivates these individuals to increase prosocial and healthy behaviors and decrease drug/alcohol use, established prevention programs may modify their approaches to include contingency management, and use it to address the staggering public health problems homeless substance-abusing MSMs face on a daily basis.

DETAILED DESCRIPTION:
Homelessness is a significant problem plaguing American cities and homeless substance abusers face increased risks. Homeless, substance abusing men who have sex with men (MSM) suffer 80% HIV seroprevalence, engage in the sex trades and resist treatment for substance abuse. For almost 30 years, the Van Ness Recovery House (VNRH) has been providing treatment services to homeless substance-abusing MSMs in Hollywood, CA. In 1994, VNRH began providing community-based HIV prevention services to non-treatment seeking homeless substance-abusing MSMs through the VNPD, its prevention division. Contingency management interventions providing positive incentives for behavior change may be particularly well suited for this disenfranchised, high-risk cohort. Specifically, voucher-based incentive therapies (VBRT) may be particularly effective since they have established potency for increasing prosocial behaviors that successfully compete with taking drugs and for reducing drug use. A randomized, controlled trial will assign 144 non-treatment seeking homeless substance-abusing MSMs at VNPD to either VBRT or control groups (72/group) for 24 weeks, with planned follow up at 7, 9 and 12 months from randomization. The VBRT group will earn vouchers in exchange for completing prosocial and healthy behaviors and/or submitting drug-negative urine and alcohol-negative breath samples. Vouchers will be redeemable for goods located in an onsite voucher store. The control group will receive feedback regarding behaviors performed and urinalysis and breath alcohol tests, but will not receive voucher points for these behaviors. We will assess the efficacy of the VBRT intervention for increasing prosocial and healthy behavior and reducing substance abuse among these non-treatment seeking homeless substance-abusing MSMs receiving services at VNPD. We will also assess the impact of VBRT on other measures of therapeutic change consistent with a harm reduction approach, including reduction of psychiatric symptoms, decreased injection drug use and high-risk sexual behavior, increased participation in prevention programming, improvement in different domains of overall functioning (medical/social/vocational), and increased readiness to change. Additionally, we will examine whether baseline participant characteristics predict VBRT outcomes. Applying VBRT to non-treatment seeking homeless substance-abusing MSMs as well as integrating VBRT into a well-established prevention program with a harm reduction philosophy are both highly innovative. Our reinforcement contingencies will also shape behavioral steps towards more complex behaviors, employing a basic operant tenet that has not received sufficient attention. Overall, our proposed research has the potential to have a significant impact on the public health of the Los Angeles homeless, gay and bisexual community. If VBRT is efficacious for motivating non-treatment seeking homeless substance-abusing MSMs in a community-based prevention program to increase prosocial and healthy behaviors and decrease drug/alcohol use, established prevention programs may modify their approaches to include contingency management, and use it to address the staggering public health problems HGMSAs face on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified, non-treatment seeking, men who have sex with men (MSM) at least 18 years of age and eligible to participate in the VNPD Men's Program. To be eligible to participate in the VNPD Men's Program, a person must report that they have sex with men (or men and women) and actively use drugs or alcohol.
* DSM-IV diagnosis of substance dependence as determined by structured clinical interview for DSM-IV (SCID) on at least one of the following substances: alcohol, marijuana, methamphetamine, cocaine, crack, MDMA (ecstasy), opiates, or dissociative anesthetics (PCP, ketamine). These substances were chosen because they are the ones commonly used by individuals contacted by the VNPD's street outreach workers.
* Ability to understand and provide written informed consent. Also see section D6.1 for consent procedures used with vulnerable populations.
* Able to provide sufficient locator information for follow-up and/or known to VNPD outreach workers.

Exclusion Criteria: Psychiatric health issues requiring a higher level of care.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2005-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy J Reback, Ph.D., Principal Investigator — Friends Research Institute, Inc.; Jesse B Fletcher, Ph.D., Study Director — Friends Research Institute, Inc.
Locations (1):
- Friends Community Center, Los Angeles, California, United States

REFERENCES:
- [Result] Reback CJ, Peck JA, Dierst-Davies R, Nuno M, Kamien JB, Amass L. Contingency management among homeless, out-of-treatment men who have sex with men. J Subst Abuse Treat. 2010 Oct;39(3):255-63. doi: 10.1016/j.jsat.2010.06.007. Epub 2010 Jul 29. PMID 20667681
- [Result] Reback CJ, Peck JA, Fletcher JB, Nuno M, Dierst-Davies R. Lifetime substance use and HIV sexual risk behaviors predict treatment response to contingency management among homeless, substance-dependent MSM. J Psychoactive Drugs. 2012 Apr-Jun;44(2):166-72. doi: 10.1080/02791072.2012.684633. PMID 22880545
- [Result] Dierst-Davies R, Reback CJ, Peck JA, Nuno M, Kamien JB, Amass L. Delay-discounting among homeless, out-of-treatment, substance-dependent men who have sex with men. Am J Drug Alcohol Abuse. 2011 Mar;37(2):93-7. doi: 10.3109/00952990.2010.540278. Epub 2010 Dec 6. PMID 21128876
- [Derived] Fletcher JB, Reback CJ. Mental health disorders among homeless, substance-dependent men who have sex with men. Drug Alcohol Rev. 2017 Jul;36(4):555-559. doi: 10.1111/dar.12446. Epub 2016 Aug 12. PMID 27516073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from April 2005 through Feb 2008 via flyers posted throughout the community, and word of mouth.
Period: Overall Study
Arm/Group | Control | Contingency Management
Started | 67 | 64
Completed | 67 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Contingency Management | Total
Number analyzed (Participants) | 67 | 64 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 64 | 131
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.5 (8.7) | 36.3 (8.7) | 36.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 67 | 64 | 131
Region of Enrollment [Number; unit: participants]
  United States | 67 | 64 | 131

OUTCOME MEASURES:

1. Primary Outcome: Amount ($) Earned for Targeted Prosocial and Healthy Behaviors
Description: Participants earned contingency management vouchers for targeted prosocial and healthy behaviors. 1 voucher = $1
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: $ Vouchers
Arm/Group | Control | Contingency Management
Number analyzed (Participants) | 0 | 64
$ Vouchers |  | 16.21 (11.85)

2. Primary Outcome: Proportion of Level 1 (i.e., Drug Negative Urines and Alcohol Negative Breath) Clean Urine Samples Provided at 12-month Follow-up, by Condition.
Time Frame: 24 Weeks
Measure: Number; unit: Proportion of Lvl 1 Clean Urine Samples
Arm/Group | Control | Contingency Management
Number analyzed (Participants) | 67 | 64
Proportion of Lvl 1 Clean Urine Samples | 0.36 | 0.61

3. Secondary Outcome: Self-reported Psychiatric Symptoms at 12-month Follow-up.
Description: As measured by the General Severity Index (GSI), a summary domain included on the Brief Symptom Inventory. The GSI combines information on both the number of symptoms described and the severity of those symptoms. Lower values on the GSI indicate less severe symptoms. Normative non-patient populations have been shown to have average GSI scores with a mean of 0.30 and a standard deviation of 0.31. Normative outpatient psychiatric patients have demonstrated GSI scores with a mean of 1.32 with a standard deviation of 0.72.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Units of General Severity Index
Arm/Group | Control | Contingency Management
Number analyzed (Participants) | 67 | 64
Units of General Severity Index | 1.01 (0.78) | 0.60 (0.62)

4. Secondary Outcome: Self-reported Sexual Behaviors at 12-month Follow-up
Description: Count of recent (past 30 days) male sexual partners.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Sexual Partners
Arm/Group | Control | Contingency Management
Number analyzed (Participants) | 67 | 64
Sexual Partners | 3.33 (9.7) | 0.70 (1.1)

ADVERSE EVENTS:
Arm/Group | Control | Contingency Management
Serious Adverse Events (participants affected / at risk) | 2/67 | 1/64
Other Adverse Events (participants affected / at risk) | 0/67 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=67) | Contingency Management (N=64)
Gall Bladder Surgery (Surgical and medical procedures) | 1 (1) | 0 (0) — Participant had gall bladder surgery for reasons unrelated to the study protocol.
Sprained Ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Hospitalized for two weeks due to a sprained ankle. Deemed unrelated to the protocol.
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) — Deemed unrelated to the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No